CLINICAL TRIAL: NCT06929650
Title: Thermo-Ablation With Radiofrequency Medical Technologies to Treat Thyroid Cancers
Brief Title: The Safety and Feasibility of Radiofrequency Ablation to Treat Low-risk Thyroid Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jesse Pasternak, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-5788
Record Dates: First submitted 2025-03-31; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Nodule; Thyroid Cancer
Keywords: Radiofrequency Ablation; Feasibility; Adverse Event; Thyroid nodule
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants receive RFA intervention for thyroid nodule.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency energy is delivered to the thyroid nodule via the medical device. This device is a system consisting of 3 main components:
  1. VIVA combo RF system (generator and pump)
  2. single foot switch
  3. electrode (5mm, 7mm, 10mm, or adjustable).

SUMMARY:
The goal of this clinical trial is to test radiofrequency ablation (RFA) in thyroid cancers ≤2 cm in diameter. The main question it aims to answer is:

• What is the feasibility of RFA use for low-risk thyroid cancers (≤2 cm)?

Participants will undergo a set of pre-procedural scans of the target thyroid nodule and undergo the RFA procedure/intervention. Then, participants will partake in three follow-up appointments at 4 weeks, 6 months, and 12 months post-procedure as per standard of care.

DETAILED DESCRIPTION:
This is a single center, prospective case series designed to assess the feasibility of RFA therapy (using an investigational RFA device) in a small cohort of participants at University Health Network Toronto. We hypothesize that it will be safe and feasible to use RFA therapy at the University Health Network, Toronto. Further, we believe participants will maintain a good quality of life in the postoperative period, including most avoiding hypothyroidism.

Patients will follow the standard clinical work-up to undergo surgery (e.g. lab parameters and preoperative scans). Patients will - after written informed consent - undergo the RFA procedure.

Within the first year there will be three follow-ups with the participants at:

* 4 weeks
* 6 months
* 12 months post-procedure. After the 12-month follow-up, participants will have follow-up appointments every 6 months until the end of the study.

During these follow-up appointments, the clinician will note any complications or adverse events, and participants will undergo blood sample draws to evaluate serum thyroid stimulating hormone (TSH) concentration. Thyroid nodule size is captured at each follow-up post-procedure via ultrasound, and a re-biopsy may be performed after 12 months to determine if there is material change in the cellular type of the thyroid nodule.

Cost of RFA treatment (probes, human resources, clinic time, complications) compared to traditional thyroidectomy (instruments, human resources, operating room time, hospital stay, complications) will also be compared to historical controls for thyroidectomy costs based on past literature to evaluate the feasibility of RFA as an intervention in this population.

Patients will be given a questionnaire at baseline and post-RFA (~7-9 months) which includes the following components:

* thyroid cancer treatment status;
* the Decision Regret Scale (0 to 100) where 100 represents maximal regret (only post-RFA);
* the Fear of Progression Questionnaire- Short Form questionnaire (focused on thyroid cancer disease progression);
* the Hospital Anxiety and Depression Scale (HADS);
* the MD Anderson Symptom Inventory for thyroid cancer (MDASI-Thy), a disease-specific quality of life questionnaire; and
* the Body Image Scale (BIS), a questionnaire on body image perception for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with:

* Nodule less than or equal to 2cm in size

  a. Specifically: Bethesda 5/6
* Their age is ≥18 years and ≤100 years
* Able to provide written consent
* Able to attend required follow-ups as per the protocol

Exclusion Criteria:

* Patients <18 years old
* Pregnant women
* Any concern for invasive or metastatic thyroid cancer
* Previously treated for thyroid cancer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications | Immediately after the procedure, and 4 weeks/6 months/12 months post-procedure.
  Rate of complications, including pain, burns, recurrent laryngeal nerve palsy, hematoma, nodule rupture, and deviation from euthyroidism

SECONDARY OUTCOMES:
Effectiveness | 4 weeks/6 months/12 months post-procedure.
  Volume reduction rate of thyroid nodule (%)
Effectiveness | 4 weeks/6 months/12 months post-procedure.
  Description of overall symptoms
Effectiveness | 4 weeks/6 months/12 months post-procedure.
  Cosmesis score reduction (scale 0-10 where 0 indicates no issues with cosmesis)
Quality of life | 7-9 months post-procedure.
  The Body Image Scale is a patient-reported questionnaire used to assess how cancer or its treatment affects a person's perception of their body. It asks about feelings related to appearance, self-consciousness, and changes in how the person views their body after receiving RFA.
  Responses are given on a 4-point scale: "Not at all," "A little," "Quite a bit," and "Very much." Higher scores generally indicate greater body image concerns or distress.
Quality of life | 7-9 months post-procedure.
  The Fear of Progression Questionnaire (FoP-Q) is a validated tool used to assess a patient's anxiety or fear that their illness (thyroid cancer) may worsen or return.
  It includes questions about emotional, social, and physical concerns related to disease progression.
  Responses are rated on a 5-point scale: "Never," "Seldom," "Sometimes," "Often," and "Very often." Higher scores reflect greater fear or worry about the illness progressing.
Quality of life | 7-9 months post-procedure.
  The MD Anderson Symptom Inventory (MDASI) is a validated questionnaire used to assess the severity and impact of cancer-related symptoms on a patient's daily functioning.
  It includes core symptom items (e.g., pain, fatigue, nausea) rated on a 0-10 scale (0 = not present, 10 = as bad as you can imagine).
  It also measures how these symptoms interfere with daily life (e.g., general activity, mood, work).
Quality of life | 7-9 months post-procedure.
  The Decision Regret Scale is used to measure a patient's regret after undergoing RFA.
  It includes statements rated on a 5-point Likert scale: "Strongly agree" to "Strongly disagree." It assesses whether patients feel that choosing RFA was helpful or if they regret the decision.
  Higher scores indicate greater regret about the decision.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse D Pasternak, MD, MPH, Principal Investigator — University Health Network (UHN) Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No